CLINICAL TRIAL: NCT04211987
Title: Evaluation of Functional Rehabilitation Fast Track Total Hip Arthroplasty vs Standard Care: a Randomized Controlled Trial
Brief Title: Fast Track Total Hip Arthroplasty vs Standard Care
Acronym: FastTrack-H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-19
Record Dates: First submitted 2019-12-23; First posted 2019-12-26 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Hip Osteoarthritis; Hip Pain Chronic
Keywords: fast track care; Total Hip Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fast track care protocol (Active Comparator): patients treated using fast track care protocol
  Interventions: Procedure: fast track care protocol
- Standard care protocol (Active Comparator): patients treated using standard care protocol
  Interventions: Procedure: standard care protocol

INTERVENTIONS:
Procedure: fast track care protocol — fast track care consists in educational preoperative preparation for patients, particular strategies for controlling pain and bleeding and intensive early rehabilitation protocol.
  Arms: Fast track care protocol
Procedure: standard care protocol — standard care protocol consists in the same surgical intervention without educational preoperative preparation for patients and intensive early rehabilitation protocol.
  Arms: Standard care protocol

SUMMARY:
Fast-track total hip arthroplasty (THA) is a well-established concept including optimized logistics and evidence-based treatment, focusing on minimizing surgical stress and improved post-operative recovery. The aim of this protocol is to compare the standard care and fast track total hip arthroplasties in terms of functional and subjective outcomes, hospital staying, number of transfusions and analgesic consumption.

DETAILED DESCRIPTION:
The aim of this protocol is to compare standard care and fast track total hip arthroplasties. The fast track care consists of:

* preoperative educational lesson in which orthopedic surgeon, anesthesiologist and physiotherapist illustrate the operative and post operative path to the patients
* antalgic protocol administered only orally
* early rehabilitation care. The day of the surgical operation, the physiotherapist helps the patient reach the upright position. The standard care consists of usual antalgic and physiotherapy post-operative care:
* Antalgic protocol consist in intravenous drugs
* the first physiotherapy session is the day after surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by hip osteoarthritis, eligible for primary total hip arthroplasty
* BMI < 32
* American Society of Anesthesiologists physical status classification system (ASA) </= 2
* preoperative hemoglobin (HB) >13 g/dl
* patients eligible for spinal anesthesia
* presence of a care-giver

Exclusion Criteria:

* psychiatric diseases
* preoperative use of crutches
* ASA > 3
* preoperative HB < 13 g/dl

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Early functional outcomes | Third post operative day
  Early functional outcomes are collecting using Lowa Level of Assistance(ILOA) during the third post-operative day.
  This scale is able to provide data on the autonomy reached by the patient in the first postoperative period going to investigate five main motor activities (get up from supine to seated, from sitting to standing position, walk around, take three steps, the speed of walking). the total score can vary from 0 to 50, where 50 indicates better functional results.

SECONDARY OUTCOMES:
hospital staying | Third post operative day
  The collection of hospital stay for each patient. The fast track expecting hospital stay is three days
Harris Hip Score (HHS) | 6 weeks after surgery
  The collection of functional outcomes score HHS at 6 weeks. The HHS is a measure of dysfunction so the higher the score, the better the outcome for the individual. The maximum score possible is 100. Results can be interpreted with the following: <70 as poor result; 70-80 as fair, 80-90 as good, and 90-100 as excellent results.
  The collection of functional outcomes score HHS at 6 weeks. The HHS is a measure of dysfunction so the higher the score, the better the outcome for the individual. The maximum score possible is 100. Results can be interpreted with the following: <70 as poor result; 70-80 as fair, 80-90 as good, and 90-100 as excellent results.
  The collection of functional outcomes score HHS at 6 weeks. The HHS is a measure of dysfunction so the higher the score, the better the outcome for the individual. The maximum score possible is 100. Results can be interpreted with the following: <70 as poor result; 70-80 as fair, 80-90 as good, and 90-100 as excellent results.
Harris Hip Score (HHS) | 3 months after surgery
  The collection of functional outcomes score HHS at 3 month after surgery. The HHS is a measure of dysfunction so the higher the score, the better the outcome for the individual. The maximum score possible is 100. Results can be interpreted with the following: <70 as poor result; 70-80 as fair, 80-90 as good, and 90-100 as excellent results
Harris Hip Score (HHS) | 6 months after surgery
  The collection of functional outcomes score HHS at 6 month after surgery. The HHS is a measure of dysfunction so the higher the score, the better the outcome for the individual. The maximum score possible is 100. Results can be interpreted with the following: <70 as poor result; 70-80 as fair, 80-90 as good, and 90-100 as excellent results.
Harris Hip Score (HHS) | 12 months after surgery
  The collection of functional outcomes score HHS at 12 month after surgery. The HHS is a measure of dysfunction so the higher the score, the better the outcome for the individual. The maximum score possible is 100. Results can be interpreted with the following: <70 as poor result; 70-80 as fair, 80-90 as good, and 90-100 as excellent results.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 6 weeks after surgery
  The collection of functional outcomes score Womac at 6 weeks after surgery. The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 3 months after surgery
  The collection of functional outcomes score Womac at 3 months after surgery. The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 6 months after surgery
  The collection of functional outcomes score Womac at 6 months after surgery. The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 12 months after surgery
  The collection of functional outcomes score Womac at 12 months after surgery. The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
  The collection of functional outcomes score Womac at 12 months after surgery. The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Dante Dallari, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzli, Bologna, Italy